CLINICAL TRIAL: NCT01701921
Title: The Effects of Pregabalin on Acute and Chronic Postoperative Pain After Cardiac Surgery
Brief Title: The Effects of Pregabalin on Postoperative Pain After Cardiac Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Aikaterini Bouzia, MD, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 7/13-07-2011
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Pain
Keywords: cardiac surgery; pregabalin; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pregabalin 75 (Experimental): Pregabalin 75mg by mouth one hour before surgery
  Interventions: Drug: Pregabalin 75mg
- Pregabalin 150 (Active Comparator): Pregabalin 150mg by mouth one hour before surgery
  Interventions: Drug: pregabalin 150 mg
- Sugar pill (Placebo Comparator): Placebo : Sugar pill manufactured to mimic pregabalin capsule by mouth one hour before surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin 75mg — Pregabalin 75mg by mouth one hour before surgery
  Other Names: Lyrica
  Arms: Pregabalin 75
Drug: pregabalin 150 mg — pregabalin 150mg by mouth one hour before surgery
  Other Names: Lyrica
  Arms: Pregabalin 150
Drug: Placebo — Sugar pill designed to mimic pregabalin capsule, by mouth one hour before surgery
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether pregabalin is effective in the treatment of acute postoperative pain after cardiac surgery if administered before the surgery.

DETAILED DESCRIPTION:
Pregabalin was introduced as an antiepileptic drug with analgesic anti-hyperalgesic and anxiolytic properties and was also used to treat neuropathic pain. In recent years it has been used as part of a multimodal management of acute postoperative pain after various types of surgery. We study the effect of pregabalin administered before cardiac surgery on acute and chronic postoperative pain. Post CABG syndrome is well known since 1980 and various analgesic methods have been used from time to time (opioids, regional analgesia, non-steroidal anti-inflammatory drugs). In our research patients will be divided into three groups. The control group will receive a placebo capsule before surgery. The second group will receive 75mg of pregabalin per os before surgery while the third will receive 150mg of pregabalin. After the surgery all patients will be connected to an intravenous PCA morphine pump for 48 hours. The postoperative pain will be assessed with the Visual Analogue Scale (0-10) every day. Total morphine consumption by the patients as well as any other pain medications administered supplementary will be registered and compared between the different groups. Remaining postoperative pain will be assessed after 3 months. The results will be statistically analyzed in order to determine whether there is significant difference in pain management between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age 18-85years who are undergoing cardiac surgery

Exclusion Criteria:

* Chronic pain syndromes
* Renal failure
* Age >85
* Allergy to Pregabalin
* Patients already taking pregabalin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-07; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
opioid consumption and other analgesics after surgery | 24 hours after surgery
  Patients will be questioned about postoperative pain and opioid consumption will be measured during the first 24 hours after surgery. Other analgesics they may receive will also be recorded.

SECONDARY OUTCOMES:
Remaining surgery related pain and analgesics consumption | 3 months after surgery
  Patients will be questioned three month after surgery about the presence of post operative pain, whether it affects their quality of life and whether they are receiving pain treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aikaterini A Bouzia, Medicine, Principal Investigator — PhD candidate, School of Medicine, Univercity of Larissa; Georgios Vretzakis, Medicine, Study Director — Associate Professor of Anaesthesiology, Schooll of Medicine, University of Larissa
Locations (1):
- Univercity Hospital of Larissa, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided